CLINICAL TRIAL: NCT01346748
Title: The Role of Statins in Preventing Cerebral Vasospasm Secondary to Subarachnoid Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Eberval Gadelha Figueiredo, Neurology department of São Paulo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1268/09
Record Dates: First submitted 2011-04-27; First posted 2011-05-03 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: vasospasm prevention
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Statin (Experimental)
  Interventions: Drug: statin

INTERVENTIONS:
Drug: statin — Sinvastatin 80 mg per day - 21 days versus placebo

SUMMARY:
Delayed ischemia caused by cerebral vasospasm remains a common cause of morbidity and mortality after aneurysmal subarachnoid hemorrhage. A great deal of drugs has been tested in the last years. Phase II randomized clinical trials have demonstrated that statin decreases the incidence of symptomatic cerebral vasospasm after spontaneous subarachnoid hemorrhage. Clinical, double blind, randomized controlled trials with placebo. Discussion: Even though some articles have shown that statins provide better prognosis, some issues remain in debate, e.g., treatment duration and the choice of the statin.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old, Hunt-hess scale < 3

Exclusion Criteria:

* Liver disfunction, previous use of statin, hunt-hess scale 4 or 5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-08 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
The role of statins in preventing cerebral vasospasm secondary to subarachnoid hemorrhage | 6 months
  Diference in clinical outcome between patients who will or won't receive sinvastatin.

CONTACTS AND LOCATIONS:
Overall Officials: Eberval Figueiredo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas, São Paulo, São Paulo, Brazil